CLINICAL TRIAL: NCT04395118
Title: STOP-HCC Evidence-Based Hepatocellular Cancer Prevention Through Treatment of Hepatitis C Virus Infection
Brief Title: STOP HCC: Mailed HCV Treatment Outreach Program for HCC Prevention for Elevated LFTs
Acronym: STOP-HCC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will not be conducted as a RCT due to limited project timeline.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STU 072015-022
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis C; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients randomized to Group 1 will receive visit-based HCV screening, as offered by clinic providers as part of usual care. Providers must identify at-risk patients who are eligible for HCV screening, understand the benefits of screening in this population, and enter orders for HCV Ab testing. If the HCV antibody is abnormal, providers must order appropriate follow-up tests including HCV viral load to confirm HCV infection. Once HCV is confirmed, providers must refer the patients for fibrosis assessment and treatment evaluation. These efforts are augmented by an established best practice alert and health maintenance reminders.
- Mailed Outreach (Active Comparator): Patients randomized to Group 2 will receive low literacy, written materials about HCV screening in English and Spanish. The invitation will include patient-centered educational materials that discuss the risk of HCV in patients with elevated LFTs and the benefits and risks of HCV screening. The invitation will include a phone number to schedule the HCV antibody test. Once a potential subject is identified and randomized in Group 2, an outreach invitation will be mailed out. Shortly after the letter, a bilingual patient navigator will call to this potential subject. Patients will also receive centralized patient navigation to facilitate screening completion and appropriate test follow-up. He/she will help patients schedule HCV antibody testing and will assume responsibility for tracking results. Patients referred to the Hepatitis C clinic for treatment evaluation will receive reminder calls from trained and credentialed study staff 5-7 business days for scheduled appointments.
  Interventions: Behavioral: Mailed Outreach

INTERVENTIONS:
Behavioral: Mailed Outreach — The investigators will randomize elevated LFT patients (~12,000 patients) using a centrally maintained computer-generated list. Patients will be randomly assigned to one of two HCV screening strategies including: visit-based screening as part of usual care (Group 1) or mailed screening invitation outreach and centralized patient navigation (Group 2).
  Arms: Mailed Outreach

SUMMARY:
The investigators will conduct a randomized controlled trial comparing two strategies to promote HCV screening, follow-up testing, and treatment among Parkland patients who are 18 years or older who have elevated liver functioning test (LFT) results: in reach with electronic medical record alerts and provider education vs. combination of in reach and provider education plus mailed outreach and patient navigation.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 or older
* elevated liver functioning tests (AST or ALT >35 that are separated by at least one month)
* ≥ 1 outpatient visit during 12 months prior to randomization at Parkland
* no prior HCV screening (prior HCV antibody, viral load, or genotype).
* any active medical coverage
* speaks Spanish or English

Exclusion Criteria:

* a life expectancy less than one year including any history of metastatic cancer, and those who received a palliative care or hospice referral in the past year
* history of HCC.
* non-English or Spanish speakers
* no address or phone number on file

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Hepatitis C Screening | 6 months
  Proportion with HCV Ab or HCV VL within 6 months of randomization

SECONDARY OUTCOMES:
Hepatitis C Screening | 12 months
  Proportion with HCV Ab within 12 months of randomization
Hepatitis C Confirmation | 3 months
  Proportion with HCV Viral Load within 3 months of positive antibody result
Hepatitis C Linkage to Care | 6 months
  Proportion with clinic visit within 6 months of positive HCV Viral Load
Cost Per Patient Screened | 3 months
  The primary measure of costs will be the cost per Ab completion.
Cost Per HCV Diagnosis | 12 months
  The primary measure of costs will be the cost per-patient diagnosed with HCV.

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No